CLINICAL TRIAL: NCT02166736
Title: Instantaneous Wave-Free Ratio Versus Fractional Flow Reserve in Patients With Stable Angina Pectoris or Acute Coronary Syndrome. A Multicenter, Prospective, Randomized Controlled Clinical Trial Based on the Swedish Angiography and Angioplasty Registry (SWEDEHEART) Platform
Brief Title: Evaluation of iFR vs FFR in Stable Angina or Acute Coronary Syndrome
Acronym: iFR Swedeheart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U-2013-044
Record Dates: First submitted 2014-05-07; First posted 2014-06-18 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Angina Pectoris; Acute Myocardial Infarction
Keywords: Instantaneous wave Free Ratio; Fractional Flow Reserve
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Instantaneous wave-free ratio (iFR) (Experimental)
  Interventions: Device: iFR
- Fractional Flow Reserve (FFR) (Active Comparator)
  Interventions: Device: FFR

INTERVENTIONS:
Device: iFR — Treatment guided by Instantaneous wave-free ratio (iFR®)
  Arms: Instantaneous wave-free ratio (iFR)
Device: FFR — Intervention guided by Fractional Flow Reserve
  Arms: Fractional Flow Reserve (FFR)

SUMMARY:
Previous trials have demonstrated that the use of physiological assessment of stenosis severity using fractional flow reserve (FFR) is superior to angiographic assessment in percutaneous coronary intervention (PCI) and improves clinical outcome. Despite the clinical utility, FFR is used only in 10-15% of patients today. The main reasons for the low adoption rate of FFR are the prolonged procedural time, Adenosine related discomfort and cost associated with Adenosine.

Instantaneous Wave-Free ratio (iFR®) is a novel method to assess coronary lesions for functional significance. The main benefits of the method compared to FFR are that the measurement is instantaneous and does not require Adenosine infusion. Thus, the patient does not experience any discomfort from the measurement and procedural time could be shortened compared to when using FFR. This could potentially increase the adoption rate of physiologic assessment of coronary lesions.

The aim of this trial is to compare the clinical outcome of patients assessed by iFR® with patients assessed by FFR.

Furthermore, the trial will be conducted as a registry based randomized clinical trial (RRCT) which is a novel strategy to conduct clinical trials. The randomization will occur online in the Swedish angiography and angioplasty registry (SWEDEHEART) using a web based platform.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected stable angina pectoris or unstable angina pectoris/non-ST-segment elevation myocardial infarction (NSTEMI) who are scheduled to undergo coronary angiography, and who has an indication for physiology guided assessment of coronary lesions (usually 30-80% stenosis grade). In patients with suspected stable angina pectoris, any lesion may be assessed. In patients with unstable angina pectoris/NSTEMI, only the non-culprit lesion may be assessed.

Exclusion Criteria:

* Inability to provide informed consent
* Age below 18 years
* Previous randomization in the iFR-SWEDEHEART trial
* Known terminal disease with a life expectancy of less than one year.
* In patients with multi-vessel disease and other indication than stable angina pectoris, difficulty in assessing which the culprit lesion is.
* Patient with unstable hemodynamics (Killip class III-IV)
* Inability to tolerate Adenosine
* Previous Coronary artery bypass graft (CABG) with patent grafts to the interrogated vessel.
* Heavily calcified or tortuous vessel where inability to cross the lesion with a pressure wire is expected.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2037 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
All cause death, non-fatal Myocardial infarction (MI), Unplanned revascularization | 12 months

SECONDARY OUTCOMES:
All cause death | 1-5 years
Non-fatal MI | 1-5 years
Unplanned revascularization | 1-5 years
Target lesion revascularization | 1-5 years
Time to acute coronary occlusion, stent thrombosis and restenosis in treated lesions as reported in Swedish Coronary Angiography and Angioplasty Registry (SCAAR) | 1-5 years
Change in physician´s treatment strategy depending on iFR/FFR information | Day 1
  Before randomization, the operators will have to record their angiographic assessment of the coronary lesions and the theoretical treatment strategy based on the angiographic information alone. After randomization and functional assessment of lesion severity, the operators will record how iFR/FFR changed the treatment strategy.
Assessment of patient discomfort during the procedure (none/mild/moderate/severe | Day 1
Procedural time | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Götberg, MD,PhD, Principal Investigator — Department of Cardiology, Skane University Hospital, Lund University, Lund, Sweden; Ole Fröbert, Prof, Study Chair — Department of Cardiology, Örebro University Hospital, Örebro, Sweden
Locations (14):
- Skejby University Hospital, Aarhus, Denmark
- Reykjavik University Hospital, Reykjavik, Iceland
- Sweden (12):
  - Sahlgrenska University Hospital, Gothenburg
  - Halmstad sjukhus, Halmstad
  - Helsingborg County Hospital, Helsingborg
  - Kalmar County Hospital, Kalmar
  - Karlstad County Hospital, Karlstad
  - Linköping University Hospital, Linköping
  - Skane University Hospital, Lund
  - Örebro University Hospital, Örebro
  - S:t Göran County Hospital, Stockholm
  - Sundsvall County Hospital, Sundsvall
  - Uppsala University Hospital, Uppsala
  - Västerås County Hospital, Västerås

REFERENCES:
- [Derived] Eftekhari A, Holck EN, Westra J, Olsen NT, Bruun NH, Jensen LO, Engstrom T, Christiansen EH. Instantaneous wave free ratio vs. fractional flow reserve and 5-year mortality: iFR SWEDEHEART and DEFINE FLAIR. Eur Heart J. 2023 Nov 1;44(41):4376-4384. doi: 10.1093/eurheartj/ehad582. PMID 37634144
- [Derived] Berntorp K, Rylance R, Yndigegn T, Koul S, Frobert O, Christiansen EH, Erlinge D, Gotberg M. Clinical Outcome of Revascularization Deferral With Instantaneous Wave-Free Ratio and Fractional Flow Reserve: A 5-Year Follow-Up Substudy From the iFR-SWEDEHEART Trial. J Am Heart Assoc. 2023 Feb 7;12(3):e028423. doi: 10.1161/JAHA.122.028423. Epub 2023 Feb 3. PMID 36734349
- [Derived] Gotberg M, Berntorp K, Rylance R, Christiansen EH, Yndigegn T, Gudmundsdottir IJ, Koul S, Sandhall L, Danielewicz M, Jakobsen L, Olsson SE, Olsson H, Omerovic E, Calais F, Lindroos P, Maeng M, Venetsanos D, James SK, Karegren A, Carlsson J, Jensen J, Karlsson AC, Erlinge D, Frobert O. 5-Year Outcomes of PCI Guided by Measurement of Instantaneous Wave-Free Ratio Versus Fractional Flow Reserve. J Am Coll Cardiol. 2022 Mar 15;79(10):965-974. doi: 10.1016/j.jacc.2021.12.030. PMID 35272801
- [Derived] Gotberg M, Christiansen EH, Gudmundsdottir IJ, Sandhall L, Danielewicz M, Jakobsen L, Olsson SE, Ohagen P, Olsson H, Omerovic E, Calais F, Lindroos P, Maeng M, Todt T, Venetsanos D, James SK, Karegren A, Nilsson M, Carlsson J, Hauer D, Jensen J, Karlsson AC, Panayi G, Erlinge D, Frobert O; iFR-SWEDEHEART Investigators. Instantaneous Wave-free Ratio versus Fractional Flow Reserve to Guide PCI. N Engl J Med. 2017 May 11;376(19):1813-1823. doi: 10.1056/NEJMoa1616540. Epub 2017 Mar 18. PMID 28317438
- [Derived] Gotberg M, Christiansen EH, Gudmundsdottir I, Sandhall L, Omerovic E, James SK, Erlinge D, Frobert O. Instantaneous Wave-Free Ratio versus Fractional Flow Reserve guided intervention (iFR-SWEDEHEART): Rationale and design of a multicenter, prospective, registry-based randomized clinical trial. Am Heart J. 2015 Nov;170(5):945-50. doi: 10.1016/j.ahj.2015.07.031. Epub 2015 Aug 15. PMID 26542503